CLINICAL TRIAL: NCT01162109
Title: Pharmaconutrients as Therapies for Critical Illness: Zinc in Severe Sepsis
Brief Title: Zinc Therapy in Critical Illness
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Renee Stapleton, Assistant Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Zinc1017; 1K23HL105654 (NIH)
Record Dates: First submitted 2010-07-08; First posted 2010-07-14 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Severe Sepsis
Keywords: Zinc; sepsis; critical illness; mechanical ventilation; ICU
MeSH Terms: conditions — Sepsis; Critical Illness | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Severe sepsis without zinc (Placebo Comparator): Mechanically ventilated patients with severe sepsis will be randomized to receive IV zinc or placebo
  Interventions: Dietary Supplement: Zinc sulfate
- Zinc in severe sepsis (Experimental): Mechanically ventilated patients with severe sepsis will be randomized to receive IV zinc or placebo
  Interventions: Dietary Supplement: Zinc sulfate
- Healthy Volunteers receiving zinc (Experimental): Cohort of healthy volunteers will receive a single dose of 500 mcg/kg IBW IV zinc and pharmacokinetics will be measured for 8 hours. PK in sepsis patients and healthy volunteers will be compared.
  Interventions: Dietary Supplement: Zinc sulfate

INTERVENTIONS:
Dietary Supplement: Zinc sulfate — A group of 10 mechanically ventilated patients with severe sepsis will be randomized to receive 500mcg/kg IBW elemental zinc (IV) or placebo. The dose will be escalated by 250mcg/kg IBW every 10 subjects to ceiling dose of 1250 mcg/kg IBW or until toxicity develops.
  A group of healthy volunteers will also receive IV zinc (as a single dose) and the PK will be compared to that in patients with sepsis.

SUMMARY:
Sepsis is a clinical syndrome often caused by a bloodstream infection that results in a common set of symptoms termed systemic inflammatory response syndrome (SIRS). Severe sepsis (sepsis with organ failure) is the leading cause of death in critically ill patients in the US. Most patients with severe sepsis need to be treated in the intensive care unit with mechanical ventilation and intravenous antibiotics. Between 30 to 50% of all severe sepsis patients die and quality of life in survivors is substantially reduced. New therapies are needed to improve clinical outcomes in patients with sepsis.

A new area of interest in the treatment of critical illness is pharmaconutrition, in which micronutrients (like zinc) are studied and administered to determine if they affect the inflammatory response or immunologic processes in critical illness. The FDA does not regulate micronutrients and does not require rigorous pharmacokinetic (the study of how a drug or nutrient is metabolized in the body) testing so it is not clear how to dose micronutrients in critically ill patients. It is also not clear if critically ill patients would metabolize these micronutrients differently than healthy people and would need different dosing levels. This is true of zinc, the focus of this research study.

Zinc is essential for normal immune function, oxidative stress response, and wound healing, and its homeostasis is tightly regulated. Zinc deficiency occurs in >10% of Americans and leads to loss of innate and adaptive immunity and increased susceptibility to infections. The symptoms of zinc deficiency are similar to many of the symptoms of SIRS and there is strong biologic rationale to suggest that the zinc deficiency seen in nearly all sepsis patients may contribute to the development of sepsis syndrome and to the "immunoparalysis" common in sepsis patients

This study has three specific aims, 1) to perform a phase I dose-finding study of intravenous zinc in mechanically ventilated patients with severe sepsis; 2) to define the pharmacokinetic of intravenous zinc in mechanically ventilated patients with severe sepsis compared to healthy controls; and 3) to investigate the impact of zinc on inflammation, immunity, and oxidant defense in patients with severe sepsis.

A total of 40 critically ill patients from the FAHC intensive care units and 15 healthy controls will be enrolled in the study. The critically ill patient population will be divided into 4 dosing groups of 10 subjects (7 randomized to zinc and 3 to saline placebo). Group 1 will receive 500mcg/kg IBW/day elemental zinc in divided doses every 8 hours. If the 50th percentile of the normal plasma zinc range (110mcg/dL) has not been achieved in all patients by 7 days and there are no safety concerns, sequential groups of patients will receive increasing doses in 250mcg increments to the ceiling dose. Groups 2 through 4 will receive 750, 1000, and 1250mcg/kgIBW/day elemental zinc, respectively. Each participant will receive the intravenous zinc or placebo for a total of 7 days unless they die or leave the ICU earlier. Pharmacokinetic testing will be obtained from 40 of the critically ill subjects and in 15 healthy controls. Additional blood will be drawn during the infusion protocol to investigate the impact of zinc on inflammation, immunity, and oxidant defense.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis
* Requiring mechanical ventilation
* 18 years or older

Exclusion Criteria:

* >36 hours since meeting severe sepsis criteria4
* Expected ICU length of stay <72 hours
* Pre-existing gastrointestinal disease*
* Post-cardiac arrest with significant anoxic brain injury
* Creatinine clearance <40mL/min*
* Taking zinc supplement during past month*
* Has received zinc supplementation while hospitalized
* Pregnant or lactating*
* AIDS with CD4<200*
* Previous bone marrow or solid organ transplant*
* Receiving TPN with added zinc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2010-09; Primary Completion 2017-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics/pharmacodynamics | Several time points over one week during critical illness

SECONDARY OUTCOMES:
Production of TNF-alpha by circulating monocytes | Study days 1, 3, and 7
Production of IL-1beta by circulating monocytes | Study days 1, 3, and 7
Production of IL-6 by circulating monocytes | Study days 1, 3, and 7
Production of IL-8 by circulating monocytes | Study days 1, 3, and 7
Plasma TNF-alpha | Study days 1, 3, and 7
Plasma IL-1beta | Study days 1, 3, and 7
Plasma IL-6 | Study days 1, 3, and 7
Plasma IL-8 | Study days 1, 3, and 7
Serum malondialdehyde (MDA) | Study days 1, 3, and 7
Serum 8-hydroxydeoxyguanine (8-OHdG) | Study days 1, 3, and 7
Neutrophil phagocytosis | Study days 1, 3, and 7

CONTACTS AND LOCATIONS:
Overall Officials: Renee D Stapleton, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States